CLINICAL TRIAL: NCT00210509
Title: AXERT® Early miGraine Intervention Study (AEGIS): Efficacy and Safety of Almotriptan Malate (AXERT®) Versus Placebo for the Acute Treatment of Migraine Headache
Brief Title: A Study of the Effectiveness and Safety of Almotriptan Versus Placebo in the Treatment of Migraine Headache
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Ortho LLC (Industry)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004714
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-04

CONDITIONS: Migraine
Keywords: aura; Migraine; pain; headache
MeSH Terms: conditions — Migraine Disorders; Epilepsy; Pain; Headache | interventions — almotriptan

INTERVENTIONS:
Drug: almotriptan malate

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of almotriptan malate (AXERT®) 12.5 milligram tablets compared with placebo for the acute treatment of migraine headache at the earliest onset of headache pain. Almotriptan malate (AXERT®) is approved for the treatment of migraine headache, with or without aura, in adults. Patients in this study will take either almotriptan or placebo oral tablets for 3 consecutive migraine headaches.

DETAILED DESCRIPTION:
Almotriptan malate (AXERT®) is approved for the treatment of migraine headache, with or without aura, in adults. This is a multicenter, randomized, double-blind, placebo-controlled, parallel group study of adult patients with a diagnosis of migraine headache, with or without aura. Patients will be randomized (like with the toss of a coin) to receive almotriptan malate (AXERT®) or placebo for the treatment of 3 consecutive qualifying migraine headaches. After screening, patients will leave the study center with blinded study medication and an electronic subject diary (Personal Digital Assistant [PDA]). Patients will self-dose with study medication as soon as headache pain of any intensity begins (that resembles their usual migraine), but no later than 1 hour after headache pain begins. Patients will use their PDAs to record assessments such as pain intensity, symptom severity and ability to function as related to the headaches. The primary hypothesis of this study is that the percentage of patients who are pain free two hours after taking study drug at the earliest onset of headache pain is greater in the almotriptan malate (AXERT®) 12.5mg group than in the placebo group and almotriptan malate (AXERT®) is generally well-tolerated.

Almotriptan malate (AXERT®) 12.5 milligrams or placebo tablets, one by mouth at the beginning of migraine pain (within 1 hour) for 3 consecutive migraine headaches

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine, with or without aura
* At least moderate pain with migraines
* Average of 2 to 6 migraines per month for past 3 months
* Duration of headache pain at least 4 hours
* Able to tell the difference between a migraine and a tension headache
* If taking a medication to prevent migraines, patients must have been taking a maintenance dose for at least 30 days before screening
* In generally good health
* If female, using birth control

Exclusion Criteria:

* Routinely experience other type of headache that might seem like a migraine headache
* An average of 15 or more headache days per month in the past 6 months
* Migraines began after age 50
* Taking > 1 medicine for preventing migraines
* Use of any drugs on list of prohibited drugs, of opioid drugs in past 7 days, of corticosteroids in the past 30 days, of an investigational drug within 30 days
* Use of non-drug treatment for migraine in past 14 days unless have used this treatment for > 14 days and plan to continue throughout study
* Overuse of medications that treat pain or nausea
* Migraine aura without headache
* Hemiplegic or basilar migraines
* Usually have vomiting with headache
* Headaches that usually occur upon waking
* Significant unstable medical disease
* Abnormal liver, kidney, blood, or ECG laboratory or test results
* Abusing drugs or alcohol
* History of a significant mental disorder
* Pregnant or breast-feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2004-11; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Effectiveness: pain free at 2 hours (defined as a decrease from severe, moderate or mild to no pain) without the use of supplemental pain medication and/or antiemetic medication up to the 2 hour timepoint

SECONDARY OUTCOMES:
Effectiveness: time to pain free post-dosing; timed assessments to achieve pain relief at 0.5, 1, 2, 4 and 24 hours post-dosing; consistency of response; migraine-associated symptoms; migraine-associated vomiting; change in functional disability

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Ortho LLC Clinical Trial, Study Director — Janssen-Ortho LLC

REFERENCES:
- [Result] Mathew NT, Finlayson G, Smith TR, Cady RK, Adelman J, Mao L, Wright P, Greenberg SJ; AEGIS Investigator Study Group. Early intervention with almotriptan: results of the AEGIS trial (AXERT Early Migraine Intervention Study). Headache. 2007 Feb;47(2):189-98. doi: 10.1111/j.1526-4610.2006.00686.x. PMID 17300358
- See also: AXERT Early Migraine Intervention Study (AEGIS) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=293&filename=CR004714_CSR.pdf